CLINICAL TRIAL: NCT05485142
Title: The Treatment Efficacy of Prolotherapy in Bladder Voiding Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taichung Armed Forces General Hospital (Other Government)
Responsible Party: Principal Investigator, Jing-Dung, SHEN, Senior Urologist, Taichung Armed Forces General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 108B01
Record Dates: First submitted 2022-07-17; First posted 2022-08-03 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Overactive Bladder; Underactive Bladder
Keywords: neural prolotherapy; detrusor underactivity; overactive bladder
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Bladder, Underactive | interventions — Prolotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- overactive bladder (Experimental): Overactive bladder
  Interventions: Procedure: prolotherapy
- Underactive bladder (Experimental): Underactive bladder
  Interventions: Procedure: prolotherapy

INTERVENTIONS:
Procedure: prolotherapy — 5% glucose 10ml local injection peripheral to posterior tibial nerve near ankle under ultrasound guidance once a week for 4 weeks.

SUMMARY:
Voiding dysfunction including overactive bladder, underactive bladder, and neuropathic bladder. Voiding dysfunction has a great impact on life quality, especially in the elderly society. The current medication for overactive bladder has limited efficacy and the patient easily to dropout the medication because of its side-effects. The underactive bladder is a new entity of voiding dysfunction, its optimal is still unknown. Sacral neuromodulation(SNM) and posterior tibial nerve stimulation(PTNS) have been applied for both overactive bladder and underactive bladder treatment and the results is promising, but the equipment of SNM or PTNS is not available in most places. Prolotherapy using glucose local injection causing inflammatory reaction to stimulate cytokine and growth factors release. Investigators combined the concepts of posterior tibial nerve stimulation and prolotherapy to treat voiding dysfunction. Investigators anticipate it maybe a new promising treatment for voiding dysfunction.

DETAILED DESCRIPTION:
Inclusion criteria:1. Adults over 20 years-old. 2. The patient who meets the diagnostic criteria of overactive bladder or underactive bladder. 3. The patient who capable to complete 3-days voiding diary and the questionnaire. Exclusion criteria: 1. The patient has severe stress urinary incontinence, severe pelvic organ prolapse, acute urinary tract infection, urolithiasis, or urinary tract malignancy. 2. The patient who has active skin disease on legs or not suitable for leg local injection. 3. Pregnant women. Method: 40 overactive bladder patients and 40 underactive bladder patients. The patients will receive 5% glucose 10ml local injection peripheral to posterior tibial nerve near ankle under ultrasound guidance once a week for 4 weeks, then the patients will be followed up once-a-month for 3 months. OverActive Bladder Symptom Score(OABSS), Core Lower Urinary Tract Symptom score(CLSS) questionnaire, 3-days voiding diary, and urine nerve growth factor are used for assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Adults over 20 years-old.
2. The patient who meets the diagnostic criteria of overactive bladder or underactive bladder.
3. The patient who capable to complete 3-days voiding diary and the questionnaire.

Exclusion Criteria:

1. Severe stress urinary incontinence or severe pelvic organ prolapse.
2. Acute urinary tract infection.
3. Active hematuria, urolithiasis, or neoplasm of urinary tract.
4. Acute skin lesion over the ankle injection site or the patient who could not tolerate ankle injection.
5. Pregnant women.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Overactive Bladder Symptom Score | Week 0
  The improvement of overactive bladder symptom score (OABSS), OABSS ranged from 0 to 15, the higher score means more severity of overactive bladder.
Overactive Bladder Symptom Score | Week1
  The improvement of overactive bladder symptom score (OABSS), OABSS ranged from 0 to 15, the higher score means more severity of overactive bladder.
Overactive Bladder Symptom Score | Week2
  The improvement of overactive bladder symptom score (OABSS), OABSS ranged from 0 to 15, the higher score means more severity of overactive bladder.
Overactive Bladder Symptom Score | Week3
  The improvement of overactive bladder symptom score (OABSS), OABSS ranged from 0 to 15, the higher score means more severity of overactive bladder.
Overactive Bladder Symptom Score | Week4
  The improvement of overactive bladder symptom score (OABSS), OABSS ranged from 0 to 15, the higher score means more severity of overactive bladder.
Overactive Bladder Symptom Score | Week8
  The improvement of overactive bladder symptom score (OABSS), OABSS ranged from 0 to 15, the higher score means more severity of overactive bladder.
Overactive Bladder Symptom Score | Week12
  The improvement of overactive bladder symptom score (OABSS), OABSS ranged from 0 to 15, the higher score means more severity of overactive bladder.
Overactive Bladder Symptom Score | Week16
  The improvement of overactive bladder symptom score (OABSS), OABSS ranged from 0 to 15, the higher score means more severity of overactive bladder.

SECONDARY OUTCOMES:
Cystometric bladder capacity | Week0
  Cystometric bladder capacity: the volume of water instilled into bladder while performing cystometry examination.
Cystometric bladder capacity | Week4
  Cystometric bladder capacity: the volume of water instilled into bladder while performing cystometry examination.
Cystometric bladder capacity | Week16
  Cystometric bladder capacity: the volume of water instilled into bladder while performing cystometry examination.

OTHER OUTCOMES:
The improvement of Patient Perception of Bladder Condition (PPBC) | Week 0
  The PPBC measures the patients' perception of their urinary (bladder) problems. Ranged from 1 to 6. The core 1 means no bother from bladder condition, higher score means more bother form bladder condition.
The improvement of Patient Perception of Bladder Condition | Week1
  The PPBC measures the patients' perception of their urinary (bladder) problems. Ranged from 1 to 6. The core 1 means no bother from bladder condition, higher score means more bother form bladder condition.
The improvement of Patient Perception of Bladder Condition | Week2
  The PPBC measures the patients' perception of their urinary (bladder) problems. Ranged from 1 to 6. The core 1 means no bother from bladder condition, higher score means more bother form bladder condition.
The improvement of Patient Perception of Bladder Condition | Week3
  The PPBC measures the patients' perception of their urinary (bladder) problems. Ranged from 1 to 6. The core 1 means no bother from bladder condition, higher score means more bother form bladder condition.
The improvement of Patient Perception of Bladder Condition | Week4
  The PPBC measures the patients' perception of their urinary (bladder) problems. Ranged from 1 to 6. The core 1 means no bother from bladder condition, higher score means more bother form bladder condition.
The improvement of Patient Perception of Bladder Condition | Week8
  The PPBC measures the patients' perception of their urinary (bladder) problems.
The improvement of Patient Perception of Bladder Condition | Week12
  The PPBC measures the patients' perception of their urinary (bladder) problems. Ranged from 1 to 6. The core 1 means no bother from bladder condition, higher score means more bother form bladder condition.
The improvement of Patient Perception of Bladder Condition | Week16
  The PPBC measures the patients' perception of their urinary (bladder) problems. Range from 1 to 6. The core 1 means no bother from bladder condition, higher score means more bother form bladder condition.

CONTACTS AND LOCATIONS:
Overall Officials: Jing-dung Shen, Principal Investigator — Taichung Armed Forces General Hospital
Locations (1):
- Taichung Armed Forces General Hospital, Taichung, Other (Non US), Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fowler CJ, Griffiths D, de Groat WC. The neural control of micturition. Nat Rev Neurosci. 2008 Jun;9(6):453-66. doi: 10.1038/nrn2401. PMID 18490916
- [Result] Gormley EA, Lightner DJ, Faraday M, Vasavada SP; American Urological Association; Society of Urodynamics, Female Pelvic Medicine. Diagnosis and treatment of overactive bladder (non-neurogenic) in adults: AUA/SUFU guideline amendment. J Urol. 2015 May;193(5):1572-80. doi: 10.1016/j.juro.2015.01.087. Epub 2015 Jan 23. PMID 25623739
- [Result] Kaptchuk TJ. Acupuncture: theory, efficacy, and practice. Ann Intern Med. 2002 Mar 5;136(5):374-83. doi: 10.7326/0003-4819-136-5-200203050-00010. PMID 11874310
- [Result] Abraham TS, Chen ML, Ma SX. TRPV1 expression in acupuncture points: response to electroacupuncture stimulation. J Chem Neuroanat. 2011 Apr;41(3):129-36. doi: 10.1016/j.jchemneu.2011.01.001. Epub 2011 Jan 20. PMID 21256210
- [Result] Chen HC, Chen MY, Hsieh CL, Wu SY, Hsu HC, Lin YW. TRPV1 is a Responding Channel for Acupuncture Manipulation in Mice Peripheral and Central Nerve System. Cell Physiol Biochem. 2018;49(5):1813-1824. doi: 10.1159/000493627. Epub 2018 Sep 19. PMID 30231245
- [Result] Zhang T, Yu J, Huang Z, Wang G, Zhang R. Electroacupuncture improves neurogenic bladder dysfunction through activation of NGF/TrkA signaling in a rat model. J Cell Biochem. 2019 Jun;120(6):9900-9905. doi: 10.1002/jcb.28272. Epub 2018 Dec 28. PMID 30592331
- [Result] Zhao Y, Zhou J, Mo Q, Wang Y, Yu J, Liu Z. Acupuncture for adults with overactive bladder: A systematic review and meta-analysis of randomized controlled trials. Medicine (Baltimore). 2018 Feb;97(8):e9838. doi: 10.1097/MD.0000000000009838. PMID 29465566
- [Result] MacDiarmid SA, Peters KM, Shobeiri SA, Wooldridge LS, Rovner ES, Leong FC, Siegel SW, Tate SB, Feagins BA. Long-term durability of percutaneous tibial nerve stimulation for the treatment of overactive bladder. J Urol. 2010 Jan;183(1):234-40. doi: 10.1016/j.juro.2009.08.160. PMID 19913821
- [Result] Sakura S, Chan VW, Ciriales R, Drasner K. The addition of 7.5% glucose does not alter the neurotoxicity of 5% lidocaine administered intrathecally in the rat. Anesthesiology. 1995 Jan;82(1):236-40. doi: 10.1097/00000542-199501000-00028. PMID 7832306
- [Result] Tsui BC, Kropelin B, Ganapathy S, Finucane B. Dextrose 5% in water: fluid medium for maintaining electrical stimulation of peripheral nerves during stimulating catheter placement. Acta Anaesthesiol Scand. 2005 Nov;49(10):1562-5. doi: 10.1111/j.1399-6576.2005.00736.x. PMID 16223407
- [Result] Tsui BCH, Kropelin B. The electrophysiological effect of dextrose 5% in water on single-shot peripheral nerve stimulation. Anesth Analg. 2005 Jun;100(6):1837-1839. doi: 10.1213/01.ANE.0000153020.84780.A5. PMID 15920223
- [Result] Wu YT, Ho TY, Chou YC, Ke MJ, Li TY, Tsai CK, Chen LC. Six-month Efficacy of Perineural Dextrose for Carpal Tunnel Syndrome: A Prospective, Randomized, Double-Blind, Controlled Trial. Mayo Clin Proc. 2017 Aug;92(8):1179-1189. doi: 10.1016/j.mayocp.2017.05.025. PMID 28778254
- [Result] Peters KM, Carrico DJ, Perez-Marrero RA, Khan AU, Wooldridge LS, Davis GL, Macdiarmid SA. Randomized trial of percutaneous tibial nerve stimulation versus Sham efficacy in the treatment of overactive bladder syndrome: results from the SUmiT trial. J Urol. 2010 Apr;183(4):1438-43. doi: 10.1016/j.juro.2009.12.036. Epub 2010 Feb 20. PMID 20171677